CLINICAL TRIAL: NCT04719286
Title: MinSafeStart - New Decision Aid Tool to Empower Women and Promote Better Treatment of Nausea and Vomiting During Pregnancy
Brief Title: MinSafeStart - Decision Aid Tool for Better Treatment of Nausea and Vomiting During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hedvig Marie Egeland Nordeng (Other)
Responsible Party: Sponsor-Investigator, Hedvig Marie Egeland Nordeng, Professor, University of Oslo
Organization: University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MinSafeStart
Record Dates: First submitted 2021-01-11; First posted 2021-01-22 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Hyperemesis Gravidarum; Emesis; Emesis Pregnancy
MeSH Terms: conditions — Hyperemesis Gravidarum; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention is the use of the MinSafeStart mobile application. The app utilizes the Pregnancy-Unique-Quantification-of-Emesis-24 (PUQE-24) scale to categorize the women's NVP severity (e.g. mild, moderate, or severe) on a daily basis, and visualizes the fluctuations over time in a graph. Each woman will have their own personal graph based on the information they put in. They will also be able to see how their symptoms are compared to an average graph. The women will get treatment advice based on their PUQE-24 scale, e.g. dietary and lifestyle advice for mild symptoms and referral to see the doctor for moderate and severe symptoms.
  Interventions: Device: MinSafeStart app
- Control group (No Intervention): Standard care.

INTERVENTIONS:
Device: MinSafeStart app — The intervention is the opportunity of using the MinSafeStart app. Women can register their NVP severity in the app by answering a few questions daily. Based on this, they will get tailored advice on NVP, and get alert when they should see a doctor.
  Arms: Intervention group

SUMMARY:
Nausea and vomiting in pregnancy (NVP) is affecting up to 70% of pregnant women. Studies have also shown that NVP may have a profound impact on pregnant women's wellbeing and that even mild NVP symptoms have been shown to significantly reduce pregnant women's quality of life. However, NVP symptoms often occur during the first period of pregnancy where antenatal care not yet have been established.

The objective of this project is to evaluate whether the "MinSafeStart" mobile application (app) can empower pregnant women to better self-manage NVP and hence improve their quality of life.

DETAILED DESCRIPTION:
Nausea and vomiting in pregnancy (NVP) is one of the most common pregnancy-related ailments, affecting up to 70% of pregnant women. The causes of NVP are unclear but it has been described as multifactorial and complex. Studies investigating NVP and the use of antiemetics states that early recognition and treatment of the condition is important in order to prevent further deterioration. In contrary to this recommendation, many healthcare providers and pregnant women themselves are reluctant to use antiemetics due to the fear of teratogenicity. Studies have also shown that NVP may have a profound impact on pregnant women's wellbeing and that even mild NVP symptoms have been shown to significantly reduce pregnant women's quality of life. As NVP symptoms often occur during the first period of pregnancy where antenatal care not yet have been established, it is important to empower women to optimally self-manage their care to ensure maternal and fetal health.

The objective of this project is to evaluate whether the "MinSafeStart" mobile application (app) can empower pregnant women to better self-manage NVP and hence improve their quality of life.

The "MinSafeStart" app is a patient-centered app for women with NVP. The app was developed by us, in corporation with a team consisting of interaction designers, programmers, and researchers from the University Center for Information Technology (USIT) at the University of Oslo. The app utilizes the Pregnancy-Unique-Quantification-of-Emesis-24 (PUQE-24) scale to categorize the women's NVP severity (e.g. mild, moderate, or severe) on a daily basis, and visualizes the fluctuations over time in a graph. Each woman will have their own personal graph based on the information they put in. They will also be able to see how their symptoms are compared to an average graph. The women will get treatment advice based on their PUQE-24 scale, e.g. dietary and lifestyle advice for mild symptoms and referral to see the doctor for moderate and severe symptoms.

All pregnant women over 18 years experiencing NVP, and owners of a smartphone (iOS or Android) are eligible for inclusion. Participants will be randomized to either the intervention group (opportunity to use the app) or the control group (standard care).

Data will be collected by four questionnaires (from both groups) and through the MinSafeStart app (intervention group only). All questionnaires will be distributed to the participants by email. The first questionnaire (Q1) at enrollment (baseline) and questionnaire Q2, Q3, and Q4 at follow up, 2, 4, and 6 weeks after randomization respectively.

Data about the participants will, in addition, be collected from four national registries; The Norwegian Patient Registry, The Norwegian Prescription Database, The Medical Birth Registry of Norway, and the Municipality Patient and User Registry. These data will be linked to the self-reported data (by the unique identification number of every citizen in Norway) collected during the intervention study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women currently experiencing all degrees of NVP
* Owners of a smartphone (iOS or Android) with phone lock
* Speak and understand Norwegian

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 217 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Nausea and vomiting | between baseline (Q1) and 2 weeks from baseline (Q2)
  Nausea and vomiting measured by Pregnancy-Unique-Quantification-of-Emesis-24 (PUQE-24) scale. Units of measure: 0-15 where higher score indicates more severe NVP. Categorization: 0-15, mild: ≤6 points, moderate: 7-12 points, severe: ≥13-15 points
Nausea and vomiting | between baseline (Q1) and 4 weeks from baseline (Q3)
  Nausea and vomiting measured by Pregnancy-Unique-Quantification-of-Emesis-24 (PUQE-24) scale. Units of measure: 0-15 where higher score indicates more severe NVP. Categorization: 0-15, mild: ≤6 points, moderate: 7-12 points, severe: ≥13-15 points
Nausea and vomiting | between baseline (Q1) and 6 weeks from baseline (Q4)
  Nausea and vomiting measured by Pregnancy-Unique-Quantification-of-Emesis-24 (PUQE-24) scale. Units of measure: 0-15 where higher score indicates more severe NVP. Categorization: 0-15, mild: ≤6 points, moderate: 7-12 points, severe: ≥13-15 points

SECONDARY OUTCOMES:
Change in quality of life | between baseline (Q1) and 2 weeks from baseline (Q2)
  Quality of life measured by the Health-Related of Quality of Life for Nausea and Vomiting during Pregnancy" (NVPQOL). Score ranges from 30 to 210 points where lower scores indicate better quality of life
Change in quality of life | between baseline (Q1) and 4 weeks from baseline (Q3)
  Quality of life measured by the Health-Related of Quality of Life for Nausea and Vomiting during Pregnancy" (NVPQOL). Score ranges from 30 to 210 points where lower scores indicate better quality of life
Change in quality of life | between baseline (Q1) and 6 weeks from baseline (Q4)
  Quality of life measured by the Health-Related of Quality of Life for Nausea and Vomiting during Pregnancy" (NVPQOL). Score ranges from 30 to 210 points where lower scores indicate better quality of life
Decisional Conflict | between baseline (Q1) and 2 weeks from baseline (Q2)
  Decisional Conflict measured by Decisional Conflict Scale (DCS) questionnaire. Score ranges from 0 (no decisional conflict) to 100 (extreme high decisional conflict)
Decisional Conflict | between baseline (Q1) and 4 weeks from baseline (Q3)
  Decisional Conflict measured by Decisional Conflict Scale (DCS) questionnaire. Score ranges from 0 (no decisional conflict) to 100 (extreme high decisional conflict)
Decisional Conflict | between baseline (Q1) and 6 weeks from baseline (Q4)
  Decisional Conflict measured by Decisional Conflict Scale (DCS) questionnaire. Score ranges from 0 (no decisional conflict) to 100 (extreme high decisional conflict)
Knowledge | Up to 40 weeks. Measured at four time points. Baseline (Q1), 2 (Q2), 4 (Q3), and 6 (Q4) weeks from baseline.
  10 statements about nausea and vomiting, measured by numbers of correct answers (agree/unsure/disagree). 80% correct considered as sufficient high knowledge
Sick leave rates | Up to 40 weeks. Measured at four time points. Baseline (Q1), 2 (Q2), 4 (Q3), and 6 (Q4) weeks from baseline.
  Self-reported sick leave rate in percentage
Sick leave duration | Up to 40 weeks
  Self-reported sick leave duration in weeks among those with sick leave
Hospitalization duration | Up to 40 weeks. Measured at four time points. Baseline (Q1), 2 (Q2), 4 (Q3), and 6 (Q4) weeks from baseline.
  Self-reported hospitalization duration in days
Hospitalization duration | up to 40 weeks
  As reported in the Norwegian Patient Registry in days among those with hospitalization
Beliefs About Medication | Up to 40 weeks. Measured at four time points. Baseline (Q1), 2 (Q2), 4 (Q3), and 6 (Q4) weeks from baseline.
  Beliefs About Medication were measured by Pregnant women's Beliefs About Medications - twelve Pregnancy-Specific Statements. Rated in "strongly agree", "agree", "uncertain", "disagree", and "strongly disagree"
Risk evaluation | Up to 40 weeks. Measured at four time points. Baseline (Q1), 2 (Q2), 4 (Q3), and 6 (Q4) weeks from baseline.
  Risk evaluation were measured by the risk evaluation scale containing 17 substances (egg, cheese, ginger, cranberry, folic acid/folate, smoking cigarettes, alcohol, X-ray, drugs for acid reflux, paracetamol, ibuprofen, antibiotics, meclizine, metoclopramide, ondansetron, thalidomide, swine flu vaccine). Women categorize the substances on a scale from 0 (not harmful) and 10 (very harmful) about how harmful they think these funds are during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Schultz, MSc, Study Chair — Department of Pharmacy, University of Oslo; Hedvig Nordeng, Principal Investigator — Department of Pharmacy, University of Oslo
Locations (1):
- Department of Pharmacy, University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available because of data protection regulation.

REFERENCES:
- [Derived] Ngo E, Truong MB, Wright D, Nordeng H. Impact of a Mobile Application for Tracking Nausea and Vomiting During Pregnancy (NVP) on NVP Symptoms, Quality of Life, and Decisional Conflict Regarding NVP Treatments: MinSafeStart Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Jul 5;10(7):e36226. doi: 10.2196/36226. PMID 35787487